CLINICAL TRIAL: NCT03296215
Title: Pattern of Admitted Cases in Respiratory Intensive Care Unit at Assiut University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Badwy, Investigator, Assiut University
Other Study IDs: Mahmoud Badwy2017
Record Dates: First submitted 2017-09-09; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: COPD Exacerbation
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patterno of admitted cases in Respiratory Intensive Care Unit at Assiut University Hospitals and Outcome
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — To determine different patterns of admission and their Outcome

SUMMARY:
Human health comprises many different states, ranging from perfect health to critical illness, so medical facilities should be able to provide medical assistance tailored to the patient's degree of disease.

The Intensive Care Unit (ICU) serves as a place for monitoring and care of patients with potentially severe physiologic instability requiring technical and/or artificial life support. The level of care in an ICU is greater than that available on the floor or Intermediate Care Unit.

Because of the utilization of expensive resources, ICUs should, in general, be reserved for those patients with reversible medical conditions who have a "reasonable prospect of substantial recovery".

About one third of hospital mortality occurs in critically ill patients in the intensive care unit. On the other hand, critically ill patients are responsible for 10 - 20 % of global hospital costs.

It is well accepted that early appropriate referral of patients to an ICU can significantly reduce early and possibly late mortality in the critically ill.At the same time improper selection of patients for ICU who block ICU beds often limits bed availability in ICUs. This in turn adversely affects the dynamics the whole hospital.

The Respiratory Intensive Care Unit (RICU) is an area that provides closed monitoring and intensive treatment for patients with acute or exacerbated respiratory failure caused by a disease that is primarily respiratory.

ELIGIBILITY:
Inclusion Criteria:

Patients with the following conditions are candidates for admission to the respiratory Intensive Care Unit. The following conditions include, but are not limited to:

1. Acute respiratory failure requiring ventilatory support
2. Acute pulmonary embolism with haemodynamic instability
3. Massive haemoptysis
4. Upper airway obstruction

Exclusion Criteria:

Patients who are generally not appropriate for respiratory ICU admission:

1. Irreversible brain damage
2. End stage cardiac, respiratory and liver disease with no options for transplant
3. Metastatic cancer unresponsive to chemotherapy and/or radiotherapy
4. Patients with non-traumatic coma leading to a persistent vegetative state (7,8,9,10)

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only patients admitted to repiratory ICU
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
The purpose of study is determine prognosis of patients admitted in Respiratory Intensive Care Unit at Assiut University Hospitals. | First 24hours of admission.
  Assessment of Acute Physiology and Health Evaluation II (APHCHE II) score of each admitted case.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Badwy, Resident, Principal Investigator — Assiut University; Yousef Ahmad, Prof, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available for primary Outcome
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months from study completion
Access Criteria: Data access will be reviewed by internal independent review panel

REFERENCES:
- [Background] Kahn JM, Goss CH, Heagerty PJ, Kramer AA, O'Brien CR, Rubenfeld GD. Hospital volume and the outcomes of mechanical ventilation. N Engl J Med. 2006 Jul 6;355(1):41-50. doi: 10.1056/NEJMsa053993. PMID 16822995